CLINICAL TRIAL: NCT07062172
Title: Lung Cancer Screening of Family Members of Patients With Mutation-Driven Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Hari Keshava, HS Assistant Clinical Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 6367; UCI 24-118 (Other: UCI CFCCC)
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer; Driver Mutation
MeSH Terms: conditions — Lung Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low Dose CT Scan of First Degree Relatives of Lung Cancer Patients (Experimental): First degree relatives of patients with lung cancer with a known driver mutation will receive a low dose CT scan of the chest to screen for lung abnormality.
  Interventions: Diagnostic Test: Low Dose CT Scan

INTERVENTIONS:
Diagnostic Test: Low Dose CT Scan — Completed once after screening and eligibility is confirmed.

SUMMARY:
This is a single-armed screening research study which screens immediate family member of lung cancer patients with a driver mutation to see if lung cancer can be inherited and whether researchers can find lung cancer early. Immediate family members of lung cancer patients will be 40-80 years old and screened using a low dose CT scan.

ELIGIBILITY:
Cohort A:

Inclusion Criteria:

* Current diagnosis of lung cancer with a driver mutation.
* Known driver mutation (e.g. via NGS, PCR, IHC, FISH, RT-PCR etc.)
* Able and willing to give informed consent.
* Able and willing to complete the screening questionnaire.

Cohort A:

Exclusion Criteria:

* There are no exclusion criteria for Cohort A.

Cohort B:

Inclusion Criteria:

* Age 40 - 80.
* Must have a first degree relative (mother, father, sibling, biological child) eligible for Cohort A. Note: Multiple first degree relatives of a Cohort A eligible participant may be approached for participation into the trial.
* Smoked < 20 pack years; a. Pack years = numbers of packs per day × number of years smoked; b. One pack year is the equivalent of smoking an average of 20 cigarettes (1 pack) per day for a year.
* Be able to undergo a low dose chest CT scan.
* If an upper respiratory infection (pneumonia, COVID19, flu, etc.) occurred in the last 3 months, this infection must have resolved by time of enrollment.
* Able and willing to provide informed consent.
* Able and willing to comply with the protocol requirements

Cohort B:

Exclusion Criteria:

* Previous history of lung cancers.
* Symptoms suggestive of presence of current lung cancer, including (but not limited to): unexplained weight loss of over 15 pounds within the last 12 months or unexplained hemoptysis.
* Pregnant at time of enrollment.
* History of any type of cancer within 5 years, with the exception of in situ carcinomas and non-melanoma skin cancers (if excised).
* Current smoker.
* Smoked ≥ 20 pack years.
* Had a chest CT scan within 1 year of study entry.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1753 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of lung cancers found | 2 years
  Determine the number of lung cancers found in low dose CT scans of first degree relatives of lung cancer patients with known driver mutations.

SECONDARY OUTCOMES:
Number of follow-up CT scans | 2 years
  Determine the number of follow-up CT scans ordered for first degree relatives of lung cancer patients with a known driver mutation after the initial low dose CT scan with findings of lung abnormalities.
Number of lung abnormalities detected | 2 years
  Determine the number of lung abnormalities found from low dose CT scan of first degree relatives of lung c. after the initial low dose CT scan with findings of lung abnormalities.
Number and type of biopsies performed | 2 years
  Determine the number and type of biopsies performed in follow up to the finding of a lung abnormalities after a low dose CT scan of first degree relatives of lung cancer patients with a known driver mutation.
Number and type of resections performed | 2 years
  Determine the number and type of resections performed in follow up to the finding of a lung abnormality after a low dose CT scan of first degree relatives of lung cancer patients with a known driver mutation.
Number of Adverse Events related to study procedures and follow-up interventions | 2 years
  Determine the number of Adverse Events, per CTCAE 5.0, related to study procedures and follow-up interventions of immediate family members of lung cancer patients with a known driver mutation with a finding of a lung abnormality from a low dose CT scan.
Stage of Lung Cancers Found | 2 years
  Determine the stages of all lung cancers found in immediate family members of lung cancer patients with a known driver mutation.

CONTACTS AND LOCATIONS:
Locations (1):
- Chao Family Comprehensive Cancer Center University of California, Irvine, Orange, California, United States